CLINICAL TRIAL: NCT03819985
Title: Prospective Trial of Hypofractionated Pre-Operative Radiation Therapy for Localized, Resectable Soft Tissue Sarcoma of the Extremity or Superficial Trunk (HYPORT-STS)
Brief Title: Shorter Course, Hypofractionated Pre-Surgery Radiation Therapy in Treating Patients With Localized, Resectable Soft Tissue Sarcoma of the Extremity of Superficial Trunk
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0616; NCI-2018-03436 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2018-0616 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Resectable Soft Tissue Sarcoma; Stage I Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IA Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IB Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage II Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage III Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IIIA Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8; Stage IIIB Soft Tissue Sarcoma of the Trunk and Extremities AJCC v8
MeSH Terms: interventions — Radiation Dose Hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (hypofractionated RT) (Experimental): Patients receive hypofractionated radiation therapy in 15 daily fractions over 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: Hypofractionated Radiation Therapy; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated RT
  Other Names: Hypofractionated Radiotherapy; Hypofractionated
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This phase II trial studies the wound complication risk of shorter course, hypofractionated pre-surgery radiation therapy in treating patients with localized soft tissue sarcoma of the extremity of superficial trunk that can be removed by surgery. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumor cells and have fewer side effects. Shorter course hypofractionated pre surgery radiation therapy may be more convenient for patients with soft tissue sarcoma than a longer course of radiation therapy, and may result in fewer complications.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine, in patients with localized, resectable soft tissue sarcoma, whether there is a non-inferior major wound complication rate for patients receiving 42.75 Gy in 15 fractions over 3 weeks compared to historical controls who received 50 Gy in conventional fractionation over 5-6 weeks.

SECONDARY OBJECTIVES:

I. To determine whether local control rates among patients treated with 42.75 Gy in 15 fractions is similar to that observed in previous studies for patients treated with 50 Gy in conventional fractionation over 5-6 weeks.

II. To determine whether patterns of local relapse, relapse free survival, overall survival, or metastatic disease free survival for patients treated with 42.75 Gy in 15 fractions are similar to previously reported studies.

III. To determine where there is a difference in pathologic response in tumor specimens treated with 42.75 Gy in 15 fractions compared to previously reported rates of hyalinization, fibrosis, or necrosis.

IV. To explore quality of life, as measured by the Functional Assessment of Cancer Therapy-General (FACT-G), financial toxicity as measured by the Comprehensive Score for financial Toxicity (COST) Instrument, and patient reported outcomes, as measured by the Toronto Extremity Salvage Score (TESS), among individuals undergoing a shorter, hypofractionated course of pre-operative radiation therapy for soft tissue sarcoma of the extremity or superficial trunk.

V. To gather subjective data on patient treatment preferences and experiences among individuals undergoing a shorter, hypofractionated course of pre-operative radiation therapy for soft tissue sarcoma of the extremity or superficial trunk.

OUTLINE:

Patients receive hypofractionated radiation therapy in 15 daily fractions over 3 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3-4 months for 2 years, every 6 months for 3 years, and then every year for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Tumor located in the soft tissues of the extremities or superficial trunk
* Deemed a candidate for complete macroscopic resection of the primary sarcoma
* Histologically confirmed sarcoma arising in soft tissue
* Patient may have had excisional biopsy of all gross disease at an outside facility with positive or uncertain resection margins and still be eligible if the evaluating sarcoma surgeon in the participating institution recommends oncologic re-resection of the surgical bed to obtain negative margins after a course of neoadjuvant irradiation (a sandwich approach of marginal excision-->radiation therapy(RT)--> wide excision, as per our standard practice)
* No evidence of nodal or distant metastases as determined by clinical examination or any form of imaging
* Has provided written informed consent for participation in this trial
* Eastern Cooperative Oncology Group (ECOG) performance status of 3 or less
* Life expectancy greater than 6 months
* Patients capable of childbearing are using adequate contraception
* Available for follow-up

Exclusion Criteria:

* Previous radiation therapy to the site of the sarcoma or area surrounding it such that it would be encompassed by the radiation field needed to treat the current sarcoma. In other words, treatment on this trial would require re-irradiation of tissues
* Patients with nodal or distant metastases
* Women who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2027-08-31 (Estimated); Study Completion 2027-08-31 (Estimated)

PRIMARY OUTCOMES:
Time to a major wound complication (MWC) | Up to 120 days after surgery
  A Bayesian approach for the analysis of a stopping rule of higher acute wound complications for the new dose (E) will be employed.

SECONDARY OUTCOMES:
Local recurrence free survival | Up to 10 years after radiation therapy
  The data from long-term follow-up will be analyzed for the local recurrence free survival. Kaplan-Meier curves will be generated of survival estimates. We will compare these to historical controls.
Disease free survival (DFS) time | Up to 10 years after radiation therapy
  The data from long-term follow-up will be analyzed for disease-free survival. Kaplan-Meier curves will be generated of survival estimates. Will compare these to historical controls.
Time to relapse | Up to 10 years after radiation therapy
Disease specific survival time | Up to 10 years after radiation therapy
  Kaplan-Meier curves will be generated of survival estimates.
Pattern of local relapse (in radiation field, margin of field, out of radiation field) | Up to 10 years after radiation therapy
Incidence of acute toxicity other than MWC | Up to 120 days after radiation therapy
  Acute toxicity will be documented and rates tabulated.
Incidence of late onset toxicity | Up to 120 days after radiation therapy
  Late radiation toxicity will be documented and rates tabulated.
Functional outcomes | Up to 10 years after radiation therapy
  Limb function and overall patient quality of life/functional status will be documented according to the Musculoskeletal Tumor Society (MSTS) and Toronto Extremity Salvage Score (TESS) and Euroqol-5D (EQ5D), which will be summarized and analyzed as a continuous variable. Differences between mean scores will be tested using the Mann-Whitney test. Mean and median and their 95% confidence interval (CI) will be presented.
Quality of life | Up to 10 years after radiation therapy
  Limb function and overall patient quality of life/functional status will be documented according to the MSTS and TESS and Euroqol-5D (EQ5D), which will be summarized and analyzed as a continuous variable. Differences between mean scores will be tested using the Mann-Whitney test. Mean and median and their 95% CI will be presented.

CONTACTS AND LOCATIONS:
Overall Officials: Beverly A Guadagnolo, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Bishop AJ, Mitra D, Farooqi A, Swanson DM, Hempel C, Willis T, Pearlnath C, Wang WL, Ratan R, Somaiah N, Benjamin RS, Torres KE, Hunt KK, Scally CP, Keung EZ, Satcher RL, Bird JE, Lin PP, Moon BS, Lewis VO, Roland CL, Guadagnolo BA. Moderately hypofractionated, preoperative radiotherapy in patients with soft tissue sarcomas (HYPORT-STS): Updated local control, late toxicities, and patient-reported outcomes. Cancer. 2025 Jan 1;131(1):e35542. doi: 10.1002/cncr.35542. Epub 2024 Aug 27. PMID 39192597
- [Derived] Guadagnolo BA, Bassett RL, Mitra D, Farooqi A, Hempel C, Dorber C, Willis T, Wang WL, Ratan R, Somaiah N, Benjamin RS, Torres KE, Hunt KK, Scally CP, Keung EZ, Satcher RL, Bird JE, Lin PP, Moon BS, Lewis VO, Roland CL, Bishop AJ. Hypofractionated, 3-week, preoperative radiotherapy for patients with soft tissue sarcomas (HYPORT-STS): a single-centre, open-label, single-arm, phase 2 trial. Lancet Oncol. 2022 Dec;23(12):1547-1557. doi: 10.1016/S1470-2045(22)00638-6. Epub 2022 Nov 4. PMID 36343656
- See also: MD Anderson Cancer Center — http://www.mdanderson.org